CLINICAL TRIAL: NCT03673137
Title: Phase II/III of Randomized Controlled Clinical Research on Irreversible Electroporation Synchronous Chemotherapy for Locally Advanced Pancreatic Adenocarcinoma
Brief Title: Phase II/III of Randomized Controlled Clinical Research on IRE Synchronous Chemotherapy for LAPC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y2018-ZD-001
Record Dates: First submitted 2018-09-10; First posted 2018-09-17 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2020-05

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma
Keywords: gemcitabine; pancreatic adenocarcinoma; Irreversible electroporation; overall survival time
MeSH Terms: interventions — Electroporation; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous treatment group (Experimental): Gemcitabine was administered over 30 minutes immediately following percutaneous irreversible electroporation. Gemcitabine was then given once weekly for 2 weeks, followed by a week of rest from treatment. Subsequent cycles consisted of once weekly infusions for 3 consecutive weeks out of every 4 weeks.Treatment continued until disease progression was detected by mRECIST or there was unacceptable toxicity.
  Interventions: Device: Irreversible electroporation; Drug: Gemcitabine
- Traditional treatment group (Active Comparator): The initial gemcitabine administration was on day 7 following IRE treatment. Once weekly infusions for 3 consecutive weeks out of every 4 weeks.Treatment continued until disease progression was detected by mRECIST or there was unacceptable toxicity.
  Interventions: Device: Irreversible electroporation; Drug: Gemcitabine

INTERVENTIONS:
Device: Irreversible electroporation — During the IRE process, we employed a CT scanner and an ultrasound system to guide percutaneous insertion of the electrode probes (one main electrode and one to three standard electrodes were used per treatment). The electrode number, electrode-insertion mode and intraoperative parameters were decided upon during pretreatment planning. The IRE parameters were visually simulated in the pulse generator and set up as follows: energy was applied at 1500 V/cm for 90 ms/pulse for a total of 7-9 pulses. After an initial testing pulse train was discharged to establish the best voltage value, the remaining 80 pulses were completed in 1-2 minutes. After ablation, we confirmed completion of IRE by measuring real-time resistance or current changes, in addition to intraoperative ultrasound and CT.
Drug: Gemcitabine — Gemcitabine hydrochloride (Qilu pharmaceutical [Hainan] Co., Ltd. Haikou, China] was administered by intravenous infusion at a dose of 1000 mg/m2.

SUMMARY:
Previous studies have shown that irreversible electroporation (IRE) preoperative induction chemotherapy or adjuvant chemotherapy after IRE can reduce the local recurrence rate of locally advanced pancreatic cancer (LAPC) and benefit the survival of patients. According to the technical principle of electroporation therapy (EPT), when the cell membrane is electroporated, the resistance of cell membrane decreases instantaneously, which promotes the drug to enter tumor cells and significantly increases its cytotoxicity and killing effect on tumor tissue. The purpose of study is to evaluate the safety and effectiveness of simultaneous gemcitabine administration and IRE for treating LAPC. In order to provide new ideas for the treatment of LAPC.

DETAILED DESCRIPTION:
Pancreatic cancer (PC) is a highly malignant digestive tract tumor that is projected to become the second leading cause of cancer-related deaths in both the United States and Germany by 2030. The majority of patients have locally advanced pancreatic cancer (LAPC) or metastatic pancreatic cancer (MPC) at initial diagnosis; in fact, less than 20% of newly diagnosed patients are eligible for surgical resection . The 5-year relative survival rate for PC is 8%, and for those cases diagnosed at a distant stage, the 5-year survival is 3%. For LAPC, chemotherapy, such as FOLFIRINOX (5-fluorouracil, leucovorin, irinotecan, and oxaliplatin), gemcitabine plus albumin-bound paclitaxel, or gemcitabine monotherapy, is considered first-line therapy.

However, chemotherapy has been shown to have little effect on the survival rate of those with PC, leading to the evaluation of new interventions. Recently, radiofrequency, microwave, cryoablation, and other minimally invasive therapies have been proven to be effective in the treatment of LAPC. However, these temperature-dependent ablation methods may damage peripancreatic vessels, the duodenum, and the bile and pancreatic duct, leading to high morbidity and mortality. Irreversible electroporation (IRE) is a new, nonthermal local ablation method for solid tumors. It utilizes targeted delivery of millisecond electrical pulses that induce permeabilization of cell membranes, resulting in unrecoverable nanoscale perforation and apoptotic cell death without damaging the structural components of tissues.

IRE has recently been found to have unique advantages and effectiveness in the treatment of PC. There are different proportions of exposed cells in the IRE zone and the reversible electroporation (RE) zone with a standard default electric field intensity of 1500 V per cm . In the RE zone, the permeability of the cell membranes caused by electroporation can promote the diffusion of drugs into the cells and increase cytotoxicity , which might further increase tumor treatment efficacy. Indeed, a preclinical experiment has proven that IRE may potentially reduce local recurrence by allowing increased gemcitabine tissue delivery in the RE zone.

With the above in mind, this randomized, controlled clinical trial combined systemic chemotherapy and IRE for the treatment of LAPC. The aim of this study was to assess the progression-free survival (PFS), objective response rate (ORR) and adverse events after combined therapy, with a view of achieving a more effective treatment method for LAPC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed pancreatic cancer；
* Radiologic confirmation of AJCC stage III locally advanced pancreatic cancer；
* Histological or cytological confirmation of pancreatic adenocarcinoma;
* The maximum diameter of tumor is less than 5 cm；
* Biliary drainage in patients with biliary obstruction；
* PS 0-1
* Written informed consent

Exclusion Criteria:

* Resectable pancreatic adenocarcinoma;
* The tumor invaded the duodenum or stomach through mucosa；
* History of epilepsy;
* History of cardiac disease: congestive heart failure > NYHA classification 2;
* cardiac arrhythmias requiring anti-arrhythmic therapy or pacemaker;
* Coronary artery disease and myocardial infarction occurred within 6 months before the screening；
* Uncontrolled hypertension. During screening, blood pressure should be controlled at less than 160/95 mmHg.
* Any implanted metal stent/device within the area of ablation that cannot be removed;
* Any implanted stimulation device;
* Uncontrolled infection (>grade 2 according to NCI CTCAE V4.0);
* Pregnant or lactating women. Women suspected of pregnancy should be tested for pregnancy within 7 days before treatment.
* Allergy to contrast media;
* Compromised liver function: signs of portal hypertension; INR >1.5 without use of anticoagulants; ascites;
* Any condition that is unstable or that could jeopardize the safety of the subject and their compliance in the study；
* There was a history of chemotherapy within 1 months before screening；
* There was a history of IRE, cryotherapy, microwave therapy, immunotherapy and radiotherapy for pancreatic tumors within the first three months of screening；
* Other primary tumors, except adequately treated non-melanoma skin cancer, cervical carcinoma in situ or other malignant tumors, which did not recur after 5 years of treatment;
* Infection beyond control > Level 2 (NCI-CTC3.0 version);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
  The time of patient from randomization to death caused by any cause

SECONDARY OUTCOMES:
Time to progression | 3 years
  Time from randomization to radiological progression. Definition of progression is based on the RECIST amendments. Deaths during follow-up without evidence of radiological progression are censored.
Time to local recurrence | 3 years
  Time from randomization to local radiological progression. Definition of progression is based on the RECIST amendments. Deaths during follow-up without evidence of radiological progression are censored.

OTHER OUTCOMES:
Progression-free survival | 3 years
  Composite endpoint. Time from randomization to either radiological progression or death. Patients alive and free of progression at the end of follow-up are censored.
Response rate | 3 years
  Definition of response is based on the RECIST amendments.

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, Doctor, Study Chair — Guangzhou FUDA Cancer Hospital
Locations (1):
- Institutional Review Board of Guangzhou FUDA Cancer Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No